#### MeTHOS PROTOCOL SYNOPSIS: OBSERVATIONAL STUDY

Title: Metaxa's Thromboprophylaxis program

in Oncological & Surgical patients

Short Title MeTHOS

Protocol Date: December 2018

**Study Principal Investigators** 

Spyridon Xynogalos, MD, sxyn@otenet.gr Panagiotis Manikis, MD, paniman14@gmsil.com

**Co-Investigator** 

Nikolaos Ziras, MD, zirasngr@otenet.gr

Konstantinos Ntatsis George Vorias

Sub - Investigators

**Evangelos Fergadis** 

Iovatso Hristos

**David Simeonidis** 

Orestis Sidiripoulos

Georgia Migga

Chrysa Kapsokoli

Maria Leonti

Evridiki Maslimoglou

Emmanouil Mpakalinis

#### PROTOCOL SYNOPSIS

#### Study

#### Metaxa's Thromboprophylaxis program

**Title** 

in Oncological & Surgical patients

### **Study Rationale Introduction**

Venous thromboembolism (VTE) is common in cancer patients, with the risk being 4- to 7-fold higher compared with noncancer patients. [1]. VTE is associated with increased mortality, morbidity, [2,3] and burden on health care resources. [4]. The risk of recurrence and bleeding complications are major concerns during anticoagulant therapy, as up to 9% of cancer patients with VTE develop recurrent thrombotic events, despite treatment with low-molecular-weight heparin (LMWH), [5–8]. Consequently, more effective prevention measures, especially during high-risk circumstances such as the postoperative period, may improve outcomes in these patients.

## Cancer patients undergoing surgery treatment

It has been well established that major surgery itself increases the risk of VTE even in the absence of cancer. [9]. Historical data from 1970s and 1980s using routine screening procedures reported a 37% incidence of deep vein thrombosis (DVT) following general surgery in patients with cancer, in contrast to an estimated risk of 20% in patients without cancer. [10]. However, changes in surgical techniques, use of perioperative chemotherapy, and the practice of early postoperative mobilization with increased awareness of perioperative VTE likely have altered VTE incidence over time.

The absolute VTE risk varies with the type of surgery, including site, technique (e.g., open vs. laparoscopic approach), duration of surgery, type of anesthesia, the presence of postoperative infection and immobilization, and patients' comorbidities (e.g., body mass index [BMI] and previous history of VTE). Surgeries for resection of malignant tumors are associated with a particularly high risk of VTE likely because of the extensive vascular injury from tumor invasion and dissection as well as lengthy operation time, and in some cases, residual tumor or nodal mass continues to cause venous compression and stasis. Prolonged postoperative immobility is also quite common in these patients.

The risk of thrombosis is not only increased during the immediate postoperative period but also extends at least up to 30 days or even longer after surgery. In the @RISTOS study that prospectively followed 2,373 patients who underwent surgery for cancer, 40% of symptomatic VTE occurred more than 3 weeks after surgery and 46% of deaths were due to fatal pulmonary embolism (PE). [11] The investigators of the @RISTOS study found that a previous history of VTE, anesthesia lasting 2 hours or longer, bed rest for 4 days or longer, advanced tumor stage, and age 60 years or older were significant risk factors for VTE. Similarly, in the Million Women Study, the incidence of symptomatic VTE was observed to peak at 3 weeks postoperatively for all surgeries, but the risk remained

> high up to 4 to 12 months for cancer patients.[12]. Relative to patients without cancer, the risk of VTE after surgery for cancer was 91-fold higher at 6 weeks, 53-fold at 7 to 12 weeks, and 34- fold at 4 to 12 months after surgery.

Estimated risk of venous thromboembolism associated with various types of surgery 13

| Surgical setting | Incidence of DVT, % | Incidence of PE, % |
|---|---|---|
| Major abdominal and pelvic surgery (colorectal/gynecological) | 15-40 <sup>a</sup> | 1.3-2 <sup>d</sup> |
| Major open urological surgery | 15-40 <sup>a</sup> | 0.2 <sup>e</sup> |
| Neurosurgery | 15-40 <sup>a</sup> | Insufficient data |
| Thoracic surgery | 4-14 <sup>a</sup> | 5-12 <sup>f</sup> |
| Breast surgery | 0.8-2.1 <sup>b</sup> | Insufficient data |
| Laparoscopic surgery | 1-11 <sup>c</sup> | Insufficient data |

Abbreviations: DVT, deep vein thrombosis; PE, pulmonary embolism.

#### Pharmacological Prophylaxis

**Pharmacological** Prophylaxis for cancer patients undergoing surgery

Studies in the late 1980s and early 1990s showed that pharmacological prophylaxis reduces the risk of postoperative VTE by 60% compared with no prophylaxis.[14-17]

LMWH is generally the preferred choice of anticoagulant over UFH based on its ease of administration (once daily vs. twice to three times per day for UFH) and lower risk of heparin-induced thrombocytopenia (HIT).

Cancer patients may also tolerate higher doses of LMWH without increasing the bleeding risk further.[18]

The optimal duration of thromboprophylaxis after cancer surgery has not been established and the available data are limited to major abdominal and pelvic surgery. Although studies have shown that a longer duration of prophylaxis up to 1 month after major abdominal and pelvic surgery can further reduce the risk of VTE compared with standard duration (typically while in hospital or up to 7–10 days) [19-21]

In the ENOXACAN II trial, patients who received extended thromboprophylaxis (ETP) with LMWH up to 30 days after open surgery for abdominal and pelvic cancer had a 60% VTE risk reduction (95% CI: 10–82%), compared with those who received standard duration of 6 to 10 days (4.8 vs. 12%; p = 0.02).[19]

These findings are supported by a recent meta-analysis of seven RCTs and prospective studies which concluded that ETP is associated with a significant risk reduction of all VTE (2.6 vs. 5.6%; (RR: 0.44, 95% CI:

Source: Adapted and modified from Geerts et al.

<sup>&</sup>lt;sup>a</sup>Routine screening of asymptomatic patients without prophylaxis.

Symptomatic patients without prophylaxis or mechanical prophylaxis alone (from retrospective studies)

Routine screening of asymptomatic patients with or without prophylaxis.

<sup>&</sup>lt;sup>d</sup>Symptomatic patients without prophylaxis.

<sup>e</sup>Symptomatic patients without prophylaxis or mechanical prophylaxis alone.

Routine screening of asymptomatic patients with CT chest.

0.28–0.70) and proximal DVT (1.4 vs. 2.8%; RR: 0.46, 95% CI: 0.23–0.91). [22]

## Consensus guidelines on primary thromboprophylaxis in cancer patients undergoing surgery

Guidelines for thromboprophylax is for cancer patients undergoing surgery

| Methods Guideline Recommendations | | Recommendations |
|---|---|---|
| Pharmacological<br>thromboprophylaxis | ACCP 2012 | For general and abdominal-pelvic surgery and thoracic patients at high risk for VTE who are not at high risk for major bleeding complications, pharmacological prophylaxis with LMWH or LDUH is recommended over no prophylaxis. For craniotomy and spinal surgery patients at high risk for VTE, pharmacological prophylaxis should be added to mechanical prophylaxis once adequate hemostasis is established and risk of bleeding decreases |
| | ASCO 2015 | All patients with malignant disease undergoing major surgical intervention should be considered for pharmacological thromboprophylaxis with either UFH or LMWH unless contraindicated Prophylaxis should be commenced preoperatively |
| | ESMO 2011 | <ul> <li>In cancer patients undergoing major cancer surgery (laparotomy, laparoscopy,<br/>thoracotomy, or thoracoscopy lasting more than 30 min), prophylaxis with LMWHs<br/>or UFH is recommended</li> </ul> |
| thromboprophylaxis | ACCP 2012 | Mechanical prophylaxis with elastic stockings or IPC should be added to pharmacological prophylaxis in patient with high risk of VTE For high VTE risk general and abdominal pelvic surgery patients, who are also at high risk for major bleeding complications, mechanical prophylaxis, preferably with IPC, is suggested over no prophylaxis until the risk of bleeding diminishes and pharmacologic prophylaxis may be initiated For high VTE risk patients in whom the consequence of bleeding might be severe, mechanical prophylaxis is suggested over no prophylaxis |
| | ASCO 2015 | A combined regimen of pharmacological and mechanical prophylaxis may improve efficacy, especially in the highest risk patients Mechanical prophylaxis should not be used as monotherapy unless pharmacological methods are contraindicated |
| | ESMO 2011 | Mechanical methods such as pneumatic calf compression may be added to<br>pharmacological prophylaxis but should not be used as monotherapy unless<br>pharmacological prophylaxis is contraindicated because of active bleeding |
| IVC filter | ACCP 2012 | IVC filter should not be used for primary VTE prevention for all risk groups |
| | ASCO 2015 | Not specified in primary prophylaxis setting |
| | ESMO 2011 | Not specified in primary prophylaxis setting |
| Duration of<br>thromboprophylaxis | ACCP 2012 | Not specified |
| | ASCO 2015 | • 7–10 d |
| | ESMO 2011 | At least 10 d |
| Extended<br>thromboprophylaxis | ACCP 2011 | For high-risk patients undergoing abdominal or pelvic surgery for cancer who are<br>not otherwise at high risk for major bleeding complications, extended duration<br>pharmacologic prophylaxis (4 wk) with LMWH is recommended over limited-<br>duration prophylaxis |
| | ASCO 2015 | Extended prophylaxis with LMWH for up to 4 wk postoperatively should be considered for patients undergoing major abdominal or pelvic surgery for cancer who have high-risk features such as restricted mobility, obesity, history of VTE, or with additional risk factors |
| | ESMO 2011 | Cancer patients undergoing elective major abdominal or pelvic surgery should<br>receive in-hospital and postdischarge prophylaxis with LMWH for up to 1 mo after<br>surgery |

Abbreviations: IVC filter, inferior vena cava filter; LDUH, low-dose unfractionated heparin; LMWH, low-molecular-weight heparin; UFH, unfractionated heparin; VTE, venous thromboembolism.



# Introduction for cancer patients undergoing chemotherapy

Venous Thromboembolism (VTE) is a frequent malignancy complication which often results in serious health deterioration and death. The risk of deep vein thrombosis (DVT) and pulmonary embolism (PE) is considerably higher in cancer patients, compared to general population four to seven times [23, 24]. Venous thromboembolism is the second leading cause of death in patients with cancer and overall mortality is increased among patients who have both conditions. [25, 26, 27]

Evidences suggest that Thromboembolism risk could be cancer related, patient related or treatment related. This risk is highest for patients with certain types of solid tumors (stomach, pancreas, lung, gynecologic, bladder, testicular) and hematologic cancers and is increased for patients who are receiving chemotherapy 6.5 times [28] or radiotherapy, who have undergone operative procedures, who have metastatic disease, or who have inherited thrombophilias. Studies have indicated that the mechanisms of this effect may include mucin production by tumors, exposure of tissue factor rich surfaces and tissue factor bearing microparticles, cysteine proteinase production leading to thrombin generation, and local hypoxia. [28,29,30]

The development of VTE in cancer patients is associated with several adverse consequences including worsened short- and long-term prognosis and survival, mortality, morbidity, chemotherapy postponement, potential hospitalization, need for long-term anticoagulation with attendant bleeding complications and high rates of recurrent VTE [31,32]. In addition, VTE leads to significant consumption of health care resources; [33]. Therefore the optimal prevention and treatment of VTE are crucial components of patient care in this population. Currently, Low!Molecular! Weight Heparin (LMWH), is the gold standard for the CAT management for the last 15 years [34-36]

Moreover, in a variety of high-risk thrombosis clinical settings, LMWHs agents are safe and effective in preventing VTE [37-38]. Multiple randomized trials of thromboprophylaxis have been conducted focusing on ambulatory cancer patients receiving chemotherapy [39-40]. ESMO and ASCO current guidelines suggest considering thromboprophylaxis in high-risk ambulatory cancer patients with LMWHs.

Several contemporary studies have investigated independent predictors for VTEs in patients actively receiving chemotherapy leading to the development of risk models for identifying patients at highest risk. [41] The Khorana model is a validated scoring system that utilizes specific patient characteristics and laboratory values to stratify patients into low, intermediate, or high risk for venous thromboembolism;

Moreover, chemotherapy and thrombosis for over three decades, it remains an underappreciated risk that has not been routinely incorporated into thrombosis risk assessment models.[42]. Cytotoxic chemotherapy has a multifactorial contribution to the risk of thrombosis. It induces vascular injury through apoptosis. In the case of cisplatin, this leads to release of prothrombotic particles that trigger thrombin generation via tissue factor independent mechanisms along with drastically increased vWF activity. Other agents, like 5-FU, also drive thrombin formation in combination with depleted protein C activity. L-asparaginase administration is tied to drastically decreased protein C, protein S, and antithrombin levels, creating a prothrombotic milieu through loss of anticoagulant factors. VEGF inhibition does not directly lead to thrombosis, but instead 'primes' the endothelium through a VEGF starved state to be more susceptible to injury. Additionally, platelet activation through PAR-1 and increased Gp llb/llla activity in the case of immunomodulatory agents or increased vWF among others in the case of small molecule inhibitors contributes to this 'primed' state.[43-81]

Cancer patients undergoing systemic treatment for their malignancy are among the highest risk populations for thromboembolic complications; often, the treatment itself contributes to this risk. Recognition of the antineoplastic agents most likely to cause thrombosis can help raise provider awareness and lead to earlier diagnosis and treatment.

In our approach, we will protect our patient taking under consideration their treatment (surgery either chemotherapy)

#### **Study Objective**

In this study we will collect Real World Data of our clinical practice regarding Thromboprophylaxis in high thrombotic risk solid tumors patients undergoing surgical and /or chemotherapeutical treatment, for one year following the protocol initiation date.

- · Specifically we will focus on the following:
  - Number of thrombotic events
  - Anti-thrombotic management dosage & duration
  - Any bleedings related to anticoagulation
  - Patients' adherence and compliance

#### **Study Design**

This is a prospective, phase IV, observational, non-interventional cohort study that aims to record the daily clinical practice regarding thromboprophylaxis in high thrombotic risk cancer patients (under surgry or chemotherapy) initiated December 2018 for a year time. Patients demographic data, cancer type and stage, anticoagulant treatment dose & duration, efficacy (VTE events), safety (bleedings) and information about adherence will be collected; more than one outcomes could be recorded.

#### **Subject Completion/Withdrawal**

Subjects may withdraw from the study at any time without prejudice to their care. They may also be discontinued from the study at the discretion of the Investigator for lack of adherence to study treatment or visit schedules, AEs, or due to termination of study observation period. The Investigator may also withdraw subjects who violate the study plan, or to protect the subject for reasons of safety or for administrative reasons. It will be documented whether or not each subject completes the clinical study. If the Investigator becomes aware of any serious, related adverse events after the subject completes or withdraws from the study, they will be recorded in the source documents and on the CRF.

#### **Clinical Adverse Events**

Clinical adverse events (AEs) will be monitored throughout the study.

#### **Adverse Event Reporting**

Since the study procedures are not greater than minimal risk, SAEs are not expected. If any unanticipated problems related to the research involving risks to subjects or others happen during the course of this study (including SAEs) these will be reported in accordance with current regulations. AEs that are not serious but that are notable and could involve risks to subjects will be summarized in narrative format.

Authorized staff will perform periodic site visits to review CRFs for completeness, but will have no direct access to patient records; although they could request further information from the hospital staff. The anonymized data will be collated centrally and entered into an electronic database using double data entry where appropriate. Any discrepancies identified by electronic logic checks and will be resolved using data clarification forms sent to sites.

Ethics committee approval will be obtained where approval of a prospective non-interventional study is required. This study will be conducted in full accordance all applicable Research Policies and Procedures and all applicable laws and regulations. The investigators will perform the study in accordance with this protocol, will obtain consent, and will report unanticipated problems involving risks to subjects or others in accordance with Policies and Procedures and all regulatory

requirements. Collection, recording, and reporting of data will be accurate and will ensure the privacy, health, and welfare of research subjects during and after the study. **Subject Population Inclusion Criteria** key criteria for 1. Patients who were diagnosed with histological confirmed high thrombotic risk cancers (GI, thoracic, gynecologic and **Inclusion and Exclusion:** genitourinary) undergoing surgery 2. Age  $\geq$  18 years 3. ECOG 0-2 4. Life expectancy >6 months 5. Signed informed consent **Exclusion Criteria** 1. Patients who were not diagnosed with histological confirmed high thrombotic risk cancers (GI, thoracic, gynecologic and genitourinary) undergoing surgery 2. Age < 18 years 3. ECOG > 2 4. Life expectancy <6 months 5. Not signed informed consent **Study Duration** Each subject's participation will last from inclusion (enrolment visit) to follow up visit (if applicable; four weeks post hospital discharge) The entire study is expected to last by the end of 2019 (1) Screening: screening for eligibility, obtaining consent and administer **Study Phases** thromboprophylaxis **Screening** (2) Observation Period: monitoring subjects over treatment time Study (3) Follow-up Phase (only if applicable e.g. by the end of treatment **Treatment** period) Follow-Up • Symptomatic/Suspected vein thromboembolism, **Efficacy** including **Evaluations** pulmonary embolism and deep vein thrombosis Confirmation of symptomatic PE requires symptoms of PE and one of the following findings 1. A (new) intraluminal filling defect in (sub) segmental or more proximal branches on spiral CT scan; 2. A (new) intraluminal filling defect or an extension of an existing defect or a new sudden cut-off of vessels on the pulmonary angiogram;

- 3. A (new) considerable perfusion defect (~ 75% of a segment) with a local normal ventilation result (high-probability) on ventilation/perfusion lung scintigraphy (V/Q scan);
- 4. An inconclusive lung scan accompanied by documentation of (new) DVT in the lower extremities e.g., by compression ultrasound or venography.
- Confirmation of symptomatic DVT requires symptoms of DVT and:
- 1. A (new) noncompressible venous segment on ultrasonography
- Incidental PE with one of the following:
- 1. A (new) intra-luminal filling defect on CT scan, MRI scan, or pulmonary angiogram;
- An inconclusive lung scan accompanied by documentation of (new) DVT in the lower extremities e.g., by compression ultrasound or venography.
- Fatal PE is:
- 1. PE based on objective diagnostic testing or autopsy or
- 2. death not attributed to a documented cause and for which DVT/PE cannot be ruled out
- Incidental DVT with the following finding:

Confirmation of recurrent incidental DVT requires inconclusive or nosymptoms of DVT and:

1. A (new) noncompressible venous segment on ultrasonography

#### Safety Evaluations Major, clinically relevant non-major bleeding, and minor bleeding

Major bleeding will be defined as overt bleeding associated with: a fall in hemoglobin of 2 g/dL or more, or leading to a transfusion, or bleeding that occurs in a critical site or contributing to death.

• Bleeding in a critical area or organ such as:

Retroperitoneal

Intracranial

Intraocular

**Intraspinal** 

Intra-articular

Pericardial

Intramuscular with compartment syndrome

#### A clinically overt bleeding event

that is associated with a fall in hemoglobin of 2.0 g/dL (>1.24 mMol/L) or more, or

leading to a transfusion of  $\geq 2$  units of packed red blood cells or whole blood.

#### Bleeding contributing to death

Other clinically relevant non-major bleeding will be defined as overt bleeding not meeting the criteria for major bleeding but associated with medical intervention, unscheduled contact (visit or telephone call) with a physician, (temporary) cessation of study treatment, or associated with discomfort for the patient such as pain, or impairment of activities of daily life. All other bleeding events will be classified as minor

#### Statistical And Analytic Plan

Descriptional statistical analysis will be performed for all study data along with epidemiology methods. Continuing parameters will be presented with standards descriptional statistical measures (mean values, median values, percentages etc.) and the results will be presented accordingly into tables. For more complex correlations we will use, among other methods, chi-square tests, ANOVA and t-tests, in order to evaluate the relationships between different patient and disease characteristics, such as:

- Number of patients enrolled
- Tumor characteristics
- Co-morbidities
- Type of Surgical operation
- Type of antineoplastic treatment
- Type of thromboprophylaxis therapy
- Therapy outcomes
- Number of therapy disruptions for any reason
- Complications (AE- SAE)

and to present them, accordingly. Due to the fact that this is an observational study the results of all correlations will be carefully discussed and will be used only to assess hypotheses.

#### REFERENCES

References

Weillos

1 Heit JA, Silverstein MD, Mohr DN, Petterson TM, O'Fallon WM, Melton LJ III. Risk factors for deep vein thrombosis and pulmonary embolism: a population-based case-control study. Arch Intern Med 2000;160(06):809–815

- 2 Sørensen HT, Mellemkjaer L, Olsen JH, Baron JA. Prognosis of cancers associated with venous thromboembolism. N Engl J Med 2000;343(25):1846–1850
- 3 Khorana AA, Francis CW, Culakova E, Kuderer NM, Lyman GH. Thromboembolism is a leading cause of death in cancer patients receiving outpatient chemotherapy. J Thromb Haemost 2007; 5(03):632–634
- 4 Khorana AA, Dalal MR, Lin J, Connolly GC. Health care costs associated with venous thromboembolism in selected high-risk ambulatory patients with solid tumors undergoing chemotherapy in the United States. Clinicoecon Outcomes Res 2013; 5:101–108
- 5 Trujillo-Santos J, Nieto JA, Tiberio G, et al; RIETE Registry. Predicting recurrences or major bleeding in cancer patients with venous thromboembolism. Findings from the RIETE Registry. Thromb Haemost 2008;100(03):435–439
- 6 Prandoni P, Lensing AW, Piccioli A, et al. Recurrent venous thromboembolism and bleeding complications during anticoagulant treatment in patients with cancer and venous thrombosis. Blood 2002;100(10):3484–3488
- 7 Lee AY, Levine MN, Baker RI, et al; Randomized Comparison of Low-Molecular-Weight Heparin versus Oral Anticoagulant Therapy for the Prevention of Recurrent Venous Thromboembolism in Patients with Cancer (CLOT) Investigators. Low molecular-weight heparin versus a coumarin for the prevention of recurrent venous thromboembolism in patients with cancer. N Engl J Med 2003;349(02):146–153
- 8 Carrier M, Le Gal G, Cho R, Tierney S, Rodger M, Lee AY. Dose escalation of low molecular weight heparin to manage recurrent venous thromboembolic events despite systemic anticoagulation in cancer patients. J Thromb Haemost 2009;7(05):760–765
- 9 Geerts WH, Heit JA, Clagett GP, et al. Prevention of venous thromboembolism. Chest 2001;119(1, Suppl):132S–175S
- 10 Prandoni P, Piccioli A, Girolami A. Cancer and venous thromboembolism: an overview. Haematologica 1999;84(05):437–445
- 11 Agnelli G, Bolis G, Capussotti L, et al. A clinical outcome-based prospective study on venous thromboembolism after cancer surgery: the @RISTOS project. Ann Surg 2006;243(01):89–95
- 12 Sweetland S, Green J, Liu B, et al; Million Women Study collaborators. Duration and magnitude of the postoperative risk of venous thromboembolism in middle aged women: prospective cohort study. BMJ 2009;339:b4583

12

- 13 Kay T. Htun et al., Thromboprophylaxis in Cancer Patients Undergoing Surgery, Semin Thromb Hemost 2017;43:672-681 14 Ockelford PA, Patterson J, Johns AS. A double-blind randomized placebo controlled trial of thromboprophylaxis in major elective general surgery using once daily injections of a low molecular weight heparin fragment (Fragmin). Thromb Haemost 1989; 62(04):1046-1049 15 Marassi A, Balzano G, Mari G, et al. Prevention of postoperative deep vein thrombosis in cancer patients. A randomized trial with low molecular weight heparin (CY 216). Int Surg 1993;78(02): 166-170 16 Bergqvist D, Flordal PA, Friberg B, et al. Thromboprophylaxis with a low molecular weight heparin (Tinzaparin) in emergency abdominal surgery. A double-blind multicenter trial. Vasa 1996;25(02):156–160 17 Mismetti P, Laporte S, Darmon JY, Buchmüller A, Decousus H. Metaanalysis of low molecular weight heparin in the prevention of venous thromboembolism in general surgery. Br J Surg 2001; 88(07):913-930 18 Bergqvist D, Burmark US, Flordal PA, et al. Low molecular weight heparin started before surgery as prophylaxis against deep vein thrombosis: 2500 versus 5000 XaI units in 2070 patients. Br J Surg 1995;82(04):496-501
- 19 Bergqvist D, Agnelli G, Cohen AT, et al; ENOXACAN II Investigators. Duration of prophylaxis against venous thromboembolism with enoxaparin after surgery for cancer. N Engl J Med 2002;346(13): 975–980
- 20 Rasmussen MS, Jorgensen LN, Wille-Jørgensen P, et al; FAME Investigators. Prolonged prophylaxis with dalteparin to prevent late thromboembolic complications in patients undergoing major abdominal surgery: a multicenter randomized open-label study. J Thromb Haemost 2006;4(11):2384–2390
- 21 Kakkar VV, Balibrea JL, Martínez-González J, Prandoni P; CANBESURE Study Group. Extended prophylaxis with Bemiparin for the prevention of venous thromboembolism after abdominal or pelvic surgery for cancer: the CANBESURE randomized study. J Thromb Haemost 2010;8(06):1223–1229
- 22 Fagarasanu A, Alotaibi GS, Hrimiuc R, Lee AY, Wu C. Role of extended thromboprophylaxis after abdominal and pelvic surgery in cancer patients: a systematic review and meta-analysis. Ann Surg Oncol 2016;23(05):1422–1430
- 23. Heit JA, Silverstein MD, Mohr DN, Petterson TM, O'Fallon WM, Melton LJ III. Risk factors for deep vein thrombosis and pulmonary embolism: a population based case-control study. Arch InternMed2000;160:809-15.
- 24. Blom JW, Doggen CJM, Osanto S, Rosendaal FR. Malignancies, prothrombotic mutations, and the risk of venous thrombosis. JAMA 2005;293:715-22.

13

- 25. Khorana AA, Francis CW, Culakova E, Kuderer NM, Lyman GH. Thromboembo- lism is a leading cause of death in cancer patients receiving outpatient chemotherapy J Thromb Haemost 2007;5:632-4.
- 26. Khorana, A. (2011). Risk assessment and prophylaxis for vte in cancer patients. J Natl Compr Canc Netw, pp. 789-797.
- 27. Noble S et al: Epidemiology and pathophysiology of cancerassociated thrombosis. Br J Cancer. 2010 Apr 13; 102(Suppl 1): S2–S9.
- 28. Brose K M, Lee AY. Cancer-associated thrombosis: prevention and treatment. Curr. Oncol. 2008;15(suppl 1):S58-67.
- 29. Silverstein MD, H. J. (1998). Trends in the incidence of deep vein thrombosis and pulmonary embolism: A 25-year population-based study. Arch Intern Med, pp. 585
- 30. Varki A. Trousseau's syndrome: multiple definitions and multiple mechanisms. Blood 2007;110:1723-9.
- 31. Zwicker JI, Liebman HA, Neuberg D, et al. Tumor-derived tissue factor-bearing microparticles are associated with venous thromboembolic events in malignancy. Clin Cancer Res 2009;15:6830-40. 593.
- 32. Elyamany, G. (2014). Cancer-Associated Thrombosis: An Overview. Clin Med Insights Oncol., pp. 129–137.
- 33. A.W. Lensing, A. Piccioli, E. Bernardi, P. Simioni, B. Girolami, A. Marchiori, P. Sabbion, M.H. Prins, F. Noventa, A. Girolami, Recurrent venous thromboembolism and bleeding complications during anticoagulant treatment in patients with cancer and venous thrombosis, Blood 100 (2002) 3484-3488.
- 34. A.A. Khorana, Venous thromboembolism and prognosis in cancer, Thromb. Res. 125 (2010) 490–493 S0049-3848(10).
- 35. A.A. Khorana, M.R. Dalal, J. Lin, G.C. Connolly, Health care costs associated with venous thromboembolism in selected high-risk ambulatory patients with solid tumors undergoing chemotherapy in the United States, Clinico Econ. Outcomes Res. 5 (2013) 101–108.
- 36. Tzu!Fei Wang, Ang Li, David Garcia: Managing thrombosis in cancer patients. Res Pract Thromb Haemost. 2018 Jul; 2(3): 429–438
- 37. ESMO E-Learning: Management of Cancer Associated Thrombosis https://oncologypro.esmo.org/Education-Library/ESMO-E-Learning-and-V-Learning/Management-of-Cancer-Associated-Thrombosis
- 38. 7η Έκδοση (2018) των Θεραπευτικών Πρωτοκόλλων της Εταιρείας με τίτλο: «Θεραπευτικά Πρωτόκολλα Χορήγησης Χημειοθεραπευτικών Φαρμάκων σε Ασθενείς με Νεοπλασματικά Νοσήματα».
- 39. S. Sagar, J. Massey, J.M. Sanderson, Low-dose heparin prophylaxis against fatal pulmonary embolism, Br. Med. J. 4 (1975) 257–259.
- 40. A.A. Khorana et al. / Thrombosis Research xxx (2017) xxx-xxx Please cite this article as: A.A. Khorana, et al., Dalteparin thromboprophylaxis in cancer patients at high risk for venous

thromboembolism: A randomized trial, Thromb Res (2017), <a href="http://dx.doi.org/10.1016/j.thromres.2017.01.009">http://dx.doi.org/10.1016/j.thromres.2017.01.009</a>

14

41. Khorana AA, Francis CW, Culakova E, Lyman GH. Risk factors for chemotherapy-associated venous thromboembolism in a prospective observational study. Cancer. 2005;104(12):2822–2829. [PubMed]13. Doll DC, List AF, Greco FA, Hainsworth JD, Hande KR, Johnson DH. Acute vascular ischemic events after cisplatin-based combination

Acute vascular ischemic events after cisplatin-based combination chemotherapy for germ-cell tumors of the testis. Ann Intern Med. 1986;105(1):48–51. [PubMed]

- 42. Otten HM, Mathijssen J, Cate H, et al. Symptomatic Venous Thromboembolism in Cancer Patients Treated With Chemotherapy: An Underestimated Phenomenon. Arch Intern Med. 2004;164(190) [PubMed]
- 43. Numico G, Garrone O, Dongiovanni V, et al. Prospective evaluation of major vascular events in patients with nonsmall cell lung carcinoma treated with cisplatin and gemcitabine. Cancer. 2005;103(5):994–9. doi: 10.1002/cncr.20893.. [PubMed] [CrossRef]
- 44. Czaykowski PM, Moore MJ, Tannock IF. High risk of vascular events in patients with urothelial transitional cell carcinoma treated with cisplatin based chemotherapy. J Urol. 1998;160(6 Pt 1):2021–4. [PubMed]
- 45. Cunningham D, Starling N, Rao S, et al. Capecitabine and oxaliplatin for advanced esophagogastric cancer. N Engl J Med. 2008;358(1):36–46. [PubMed]
- 46. Moore Ra, Adel N, Riedel E, et al. High incidence of thromboembolic events in patients treated with cisplatin-based chemotherapy: a large retrospective analysis. J Clin Oncol. 2011;29(25):3466–73. [PubMed]
- 47. Seng S, Liu Z, Chiu SK, et al. Risk of venous thromboembolism in patients with cancer treated with Cisplatin: a systematic review and meta-analysis. J Clin Oncol. 2012;30(35):4416–26. [PubMed]
- 48. Licciardello JT, Moake JL, Rudy CK, Karp DD, Hong WK. Elevated plasma von Willebrand factor levels and arterial occlusive complications associated with cisplatin-based chemotherapy. Oncology. 1985;42(5):296–300. [PubMed]
- 49. Lechner D, Kollars M, Gleiss A, Kyrle PA, Weltermann A. Chemotherapy-induced thrombin generation via procoagulant endothelial microparticles is independent of tissue factor activity. J Thromb Haemost. 2007;5(12):2445–52. [PubMed]
- 45. Priest JR, Ramsay NK, Steinherz PG, et al. A syndrome of thrombosis and hemorrhage complicating L-asparaginase therapy for childhood acute lymphoblastic leukemia. J Pediatr. 1982;100(6):984–9. [PubMed]
- 46. Gugliotta L, Mazzucconi MG, Leone G, et al. Incidence of thrombotic complications in adult patients with acute lymphoblastic leukaemia receiving L-asparaginase during induction therapy: a retrospective study. The GIMEMA Group. Eur J Haematol. 1992;49(2):63–6. [PubMed]

15

47. Caruso V, Iacoviello L, Di Castelnuovo A, et al. Thrombotic complications in childhood acute lymphoblastic leukemia: a meta-analysis of 17 prospective studies comprising 1752 pediatric patients. Blood. 2006;108(7):2216–22. [PubMed]

- 48. Bezeaud A, Drouet L, Leverger G, Griffin JH, Guillin MC. Effect of L-asparaginase therapy for acute lymphoblastic leukemia on plasma vitamin K-dependent coagulation factors and inhibitors. J Pediatr. 1986;108(5 Pt 1):698–701. [PubMed]
- 49. Mitchell LG, Halton JM, Vegh PA, et al. Effect of disease and chemotherapy on hemostasis in children with acute lymphoid leukemia. Am J Pediatr Hematol Oncol. 1994;16(2):120–6. [PubMed]
- 50. Mitchell L, Hoogendoorn H, Giles AR, Vegh P, Andrew M. Increased endogenous thrombin generation in children with acute lymphoblastic leukemia: risk of thrombotic complications in L'Asparaginase-induced antithrombin III deficiency. Blood. 1994;83(2):386–91. [PubMed]
- 51. Jensen SA, Sørensen JB. Risk factors and prevention of cardiotoxicity induced by 5-fluorouracil or capecitabine. Cancer Chemother Pharmacol. 2006;58(4):487–93. [PubMed]
- 52. Wacker A, Lersch C, Scherpinski U, Reindl L, Seyfarth M. High incidence of angina pectoris in patients treated with 5-fluorouracil. A planned surveillance study with 102 patients. Oncology. 2003;65(2):108-12. [PubMed]
- 53. Ang C, Kornbluth M, Thirlwell MP, Rajan RD. Capecitabine-induced cardiotoxicity: case report and review of the literature. Curr Oncol. 2010;17(1):59–63. [PMC free article] [PubMed]
- 54. Grem JL, McAtee N, Murphy RF, et al. Phase I and pharmacokinetic study of recombinant human granulocyte-macrophage colony-stimulating factor given in combination with fluorouracil plus calcium leucovorin in metastatic gastrointestinal adenocarcinoma. J Clin Oncol.

1994;12(3):560–8. [PubMed]

- 55. Tournigand C, André T, Achille E, et al. FOLFIRI followed by FOLFOX6 or the reverse sequence in advanced colorectal cancer: a randomized GERCOR study. J Clin Oncol. 2004;22(2):229–37. [PubMed] 56. Feffer SE, Carmosino LS, Fox RL. Acquired protein C deficiency in patients with breast cancer receiving cyclophosphamide, methotrexate,
- 57. Edwards RL, Klaus M, Matthews E, McCullen C, Bona RD, Rickles FR. Heparin abolishes the chemotherapy-induced increase in plasma fibrinopeptide A levels. Am J Med. 1990;89(1):25–8. [PubMed]

and 5-fluorouracil. Cancer. 1989;63(7):1303–7. [PubMed]

58. Cwikiel M, Eskilsson J, Albertsson M, Stavenow L. The influence of 5-fluorouracil and methotrexate on vascular endothelium. An experimental study using endothelial cells in the culture. Ann Oncol. 1996;7(7):731–7. [PubMed]

59. Cwikiel M, Eskilsson J, Wieslander JB, Stjernquist U, Albertsson M. The appearance of endothelium in small arteries after treatment with 5-fluorouracil. An electron microscopic study of late effects in rabbits. Scanning Microsc. 1996;10(3):805–18. discussion 819. [PubMed] 60. Nevasaari K, Heikkinen M, Taskinen PJ. Tamoxifen and thrombosis.

16

- 60. Nevasaari K, Heikkinen M, Taskinen PJ. Tamoxifen and thrombosis Lancet. 1978;2(8096):946–7. [PubMed]
- 61. Jungi WF, Alberto P, Wagenknecht L, Cavalli F, Martz G, Brunner KW. Antiestrogens: a new endocrine treatment possibility in metastasizing breast neoplasms. Experiences of the Swiss Cooperative Cancer Study Group with tamoxifen. Schweiz Med Wochenschr. 1978;108(34):1317–21. [PubMed]
- 62. Fisher B, Dignam J, Wolmark N, et al. Tamoxifen in treatment of intraductal breast cancer: National Surgical Adjuvant Breast and Bowel Project B-24 randomised controlled trial. Lancet.

1999;353(9169):1993-2000. [PubMed]

63. Fisher B, Dignam J, Bryant J, et al. Five versus more than five years of tamoxifen therapy for breast cancer patients with negative lymph nodes and estrogen receptor-positive tumors. J Natl Cancer Inst.

1996;88(21):1529–42. [PubMed]

- 64. Fisher B, Costantino J, Redmond C, et al. A randomized clinical trial evaluating tamoxifen in the treatment of patients with node-negative breast cancer who have estrogen-receptor-positive tumors. N Engl J Med. 1989;320(8):479–84. [PubMed]
- 65. Saphner T, Tormey DC, Gray R. Venous and arterial thrombosis in patients who received adjuvant therapy for breast cancer. J Clin Oncol. 1991;9(2):286–94. [PubMed]
- 66. McCaskill-Stevens W, Wilson J, Bryant J, et al. Contralateral breast cancer and thromboembolic events in African American women treated with tamoxifen. J Natl Cancer Inst. 2004;96(23):1762–9. [PubMed] 67. Hernandez RK, Sørensen HT, Pedersen L, Jacobsen J, Lash TL. Tamoxifen treatment and risk of deep venous thrombosis and pulmonary embolism: a Danish population-based cohort study. Cancer. 2009;115(19):4442–9. [PubMed]
- 68. Baum M, Budzar AU, Cuzick J, et al. Anastrozole alone or in combination with tamoxifen versus tamoxifen alone for adjuvant treatment of postmenopausal women with early breast cancer: first results of the ATAC randomised trial. Lancet. 2002;359(9324):2131–9. [PubMed]
- 69. Goss PE, Ingle JN, Martino S, et al. Randomized trial of letrozole following tamoxifen as extended adjuvant therapy in receptor-positive breast cancer: updated findings from NCIC CTG MA.17. J Natl Cancer Inst. 2005;97(17):1262–71. [PubMed]
- 70. Jakesz R, Jonat W, Gnant M, et al. Switching of postmenopausal women with endocrine-responsive early breast cancer to anastrozole after

- 2 years' adjuvant tamoxifen: combined results of ABCSG trial 8 and ARNO 95 trial. Lancet. 2005;366(9484):455–62. [PubMed]
- 71. Folkman J. Angiogenesis. Annu Rev Med. 2006;57:1–18. [PubMed]
- 72. Kabbinavar F, Hurwitz HI, Fehrenbacher L, et al. Phase II, Randomized Trial Comparing Bevacizumab plus Fluorouracil (FU)/leucovorin (LV) with FU/LV Alone in Patients with. Metastatic Colorectal Cancer. 2003:60–65. [PubMed]
- 73. Hurwitz H, Fehrenbacher L, Novotny W, et al. Bevacizumab plus Irinotecan, Fluorouracil, and Leucovorin for Metastatic Colorectal Cancer. N Engl J Med. 2004:2335–2342. [PubMed]
- 74. Kabbinavar FF, Hambleton J, Mass RD, Hurwitz HI, Bergsland E, Sarkar S. Combined Analysis of Efficacy: The Addition of Bevacizumab to Fluorouracil/leucovorin Improves Survival for Patients with. Metastatic Colorectal Cancer. 2005:3706–3712. [PubMed]
- 75. Nalluri SR, Chu D, Keresztes R, Zhu X, Wu S. Risk of venous thromboembolism with the angiogenesis inhibitor bevacizumab in cancer patients: a meta-analysis. JAMA. 2008;300:2277–2285. [PubMed]
- 76. Scappaticci FA, Skillings JR, Holden SN, et al. Arterial thromboembolic events in patients with metastatic carcinoma treated with chemotherapy and bevacizumab. J Natl Cancer Inst. 2007;99:1232–1239. [PubMed]
- 77. Zangari M, Fink LM, Elice F, Zhan F, Adcock DM, Tricot GJ. Thrombotic events in patients with cancer receiving antiangiogenesis agents. J Clin Oncol. 2009;27:4865–4873. [PubMed]
- 78. Kuenen BC. Analysis of Coagulation Cascade and Endothelial Cell Activation During Inhibition of Vascular Endothelial Growth Factor/Vascular Endothelial Growth Factor Receptor Pathway in Cancer Patients. Arterioscler Thromb Vasc Biol. 2002;22(9):1500–1505. [PubMed]
- 79. Qi WX, Min DL, Shen Z, et al. Risk of venous thromboembolic events associated with VEGFR-TKIs: a systematic review and meta-analysis. Int J Cancer. 2013;132(12):2967–74. [PubMed]
- 80. Sonpavde G, Je Y, Schutz F, et al. Venous thromboembolic events with vascular endothelial growth factor receptor tyrosine kinase inhibitors: a systematic review and meta-analysis of randomized clinical trials. Crit Rev Oncol Hematol. 2013;87(1):80–9. [PubMed]
- 81. Evans CE, Grover SP, Humphries J, et al. Antiangiogenic therapy inhibits venous thrombus resolution. Arterioscler Thromb Vasc Biol. 2014;34:565–570. [PubMed]

#### **APPENDIX**

- 1. Informed Consent Form (in Greek: ENTYHO  $\Sigma$ YFKATA $\Theta$ E $\Sigma$ H $\Sigma$  META AHO ENHMEP $\Omega$ \SigmaH)
- 2. Case Report Form (In Greek: ΕΝΤΥΠΟ ΑΝΑΦΟΡΑΣ ΠΕΡΙΣΤΑΤΙΚΟΥ)